CLINICAL TRIAL: NCT00576537
Title: Phase ll Trial of Tumor Lysate-Pulsed Dendritic Cell Immunotherapy for Patients With Atypical or Malignant, Primary or Metastatic Brain Tumors of the Central Nervous System
Brief Title: Tumor Lysate Pulsed Dendritic Cell Immunotherapy for Patients With Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, John Yu, MD, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3368
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Glioblastoma
Keywords: New/Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dendritic Cell Immunotherapy (Experimental): Patients who consent to participate in the study and receive the Dendritic Cell vaccine manufactured from their own tumor cells.
  Interventions: Biological: Dendritic Cell Immunotherapy

INTERVENTIONS:
Biological: Dendritic Cell Immunotherapy — Patients will receive four vaccines.
  Other Names: Dendritic Cell vaccine

SUMMARY:
This research is being determine whether vaccinations with your own immune cells called " dendritic cells " can activate your immune system to fight your brain tumor.

DETAILED DESCRIPTION:
To become eligible for therapy the following criteria must be fulfilled:

* No age or gender limit
* Patients with atypical malignant brain tumors.
* Must have a Karnofsky performance of at least 60%
* Hematologic studies and chemistry profiles will be within the parameters of the protocol
* Tumor specimen of adequate size to yield protein concentration, tumor lysate peptide must be generated in sufficient quantity and patient must have no prior sensitivity to the components of the dendritic cell vaccine.
* Patients are excluded if they have systemic disease, presence of acute infection, known history of autoimmune disorder and pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* No age or gender limit, though minimal weight limitations for apheresis is about 15 - 20 Kg.
* Both male and female of childbearing age entering the protocol must use a medically accepted form of birth control during the study, will be required to have a negative pregnancy test for female.
* patients with atypical malignant brain tumor will be eligible.
* Patients must have a Karnofsky performance score of at least 60%
* patients may be maintained on glucocorticoid therapy at the lowest possible dose.
* Baseline hematologic studies and chemistry profiles must meet the criteria.
* Tumor specimen of adequate size to yield protein concentration in sufficient quantity.
* Tumor-lysate peptide must be generated in sufficient quantity to pulse the APC's for vaccination.
* Patient must have no prior sensitivity to the components of the dendritic cell vaccine.
* Patient must agree to consider an autopsy in the event of death in an attempt to learn more concerning the nature of this treatment and tumor biology.
* Patient must be capable of signing IRB approved Research Consent and Release of medical Records form.

Exclusion Criteria:

* Severe pulmonary, cardiac or other systemic disease associated with an unacceptable anesthetic or operative risk.
* The presence of an acute infection requiring active treatment will be criteria for delay or exclusion.
* Patients with a known history of an autoimmune disorder.
* Inability to give informed consent.
* Pregnancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2001-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety/toxicity of subcutaneous injections of autologous dendritic cells | One year
  Cytotoxic T lymphocyte (CTL) precursor frequency

CONTACTS AND LOCATIONS:
Overall Officials: John Yu, M.D., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical center, Los Angeles, California, United States

REFERENCES:
- [Derived] Jouanneau E, Black KL, Veiga L, Cordner R, Goverdhana S, Zhai Y, Zhang XX, Panwar A, Mardiros A, Wang H, Gragg A, Zandian M, Irvin DK, Wheeler CJ. Intrinsically de-sialylated CD103(+) CD8 T cells mediate beneficial anti-glioma immune responses. Cancer Immunol Immunother. 2014 Sep;63(9):911-24. doi: 10.1007/s00262-014-1559-2. Epub 2014 Jun 4. PMID 24893855